CLINICAL TRIAL: NCT03133520
Title: Effectiveness of High Flow Oxygen Therapy in Patients With Hematologic Malignancy Acute Hypoxemic Respiratory Failure
Acronym: HFOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kursat Gundogan (Other)
Responsible Party: Sponsor-Investigator, Kursat Gundogan, Associate professor, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: November, 2016
Record Dates: First submitted 2017-04-13; First posted 2017-04-28 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Acute Hypoxemic Respiratory Failure; Hematologic Malignancy
Keywords: Respiratory failure; immuncompromise patients; high flow oxygen
MeSH Terms: conditions — Respiratory Insufficiency; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard oxygen group (No Intervention): This patient groups will receive only routine oxygen therapy. Routine oxygen therapy involves administering low-to-medium oxygen flows through a nasal cannula or mask to achieve SpO2≥95%.
- High flow oxygen therapy group (Experimental): This patients group will receive high flow oxygen therapy. High flow nasal oxygen therapy is a focus of growing attention as an alternative to standard oxygen therapy. By providing warmed and humidified gas, it allows the delivery of higher flow rates [of up to 60 L/min] via nasal cannula devices, with fraction of inspired oxygen(FiO2) values of nearly 100%.
  Interventions: Device: High flow oxygen therapy

INTERVENTIONS:
Device: High flow oxygen therapy — High-flow nasal oxygen [HFNO] therapy is a focus of growing attention as an alternative to standard oxygen therapy. By providing warmed and humidified gas, HFNO allows the delivery of higher flow rates [of up to 60 L/min] via nasal cannula devices, with fraction of inspired oxygen(FiO2) values of nearly 100%.
  Arms: High flow oxygen therapy group

SUMMARY:
Effectiveness of high flow oxygen therapy in patients with hematologic malignancy acute hypoxemic respiratory failure

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) is the leading reason for ICU admission in immunocompromised patients. Usual oxygen therapy involves administering low-to-medium oxygen flows through a nasal cannula or mask to achieve SpO2≥95%.

High-flow nasal oxygen [HFNO] therapy is a focus of growing attention as an alternative to standard oxygen therapy. By providing warmed and humidified gas, HFNO allows the delivery of higher flow rates [of up to 60 L/min] via nasal cannula devices, with fraction of inspired oxygen (FiO2) values of nearly 100%. Physiological benefits of HFNO consist of higher and constant FiO2 values, decreased work of breathing, nasopharyngeal washout leading to improved breathing-effort efficiency, and higher positive airway pressures associated with better lung recruitment.

Clinical consequences of these physiological benefits include alleviation of dyspnea and discomfort, decreases in tachypnea and signs of respiratory distress, a diminished need for intubation in patients with severe hypoxemia, and decreased mortality in unselected patients with acute hypoxemic respiratory failure However, although preliminary data establish the feasibility and safety of this technique, HFNO has never been properly evaluated in immunocompromised patients.

Thus, this project aims at demonstrating that HFNO is superior to low/medium-flow (standard) oxygen, minimizing the need for endotracheal intubation

ELIGIBILITY:
Inclusion Criteria:

* Known immunosuppression defined as haematological malignancy.
* Need for oxygen therapy defined as with oxygen free arterial blood gas examination one or more of the following: (a) PaO2/FiO2<300 mmHg (b) PaCO2≤45 mmHg (c) SaO2<92%
* Respiratory distress with a respiratory rate >22/min

Exclusion Criteria:

* Refusal of study participation
* Pregnancy or breastfeeding
* Hypercapnia with a formal indication for non-invasive mechanical ventilation (NIMV) (PaCO2 ≥ 45 mmHg)
* Patients whose clinicians have decided on NIMV (Non-Invasive Mechanical Ventilation) and IMV (Invasive Mechanical Ventilation)
* Haemodynamic instability (mean arterial pressure <65 mmHg)
* Vasopressor needs
* Awareness confusion and disorientation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Intubation rate | First seven days
  Intubation rate for each group

SECONDARY OUTCOMES:
Mortality | First 28 days
  All-cause day-28 mortality
patients comforts | First 24 hours
  Patient comfort with Visual Analogue Scale (VAS) score

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Medical School, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turkoglu M, Erdem GU, Suyani E, Sancar ME, Yalcin MM, Aygencel G, Aki Z, Sucak G. Acute respiratory distress syndrome in patients with hematological malignancies. Hematology. 2013 May;18(3):123-30. doi: 10.1179/1607845412Y.0000000038. Epub 2012 Nov 15. PMID 23321772
- [Background] Lemiale V, Mokart D, Mayaux J, Lambert J, Rabbat A, Demoule A, Azoulay E. The effects of a 2-h trial of high-flow oxygen by nasal cannula versus Venturi mask in immunocompromised patients with hypoxemic acute respiratory failure: a multicenter randomized trial. Crit Care. 2015 Nov 2;19:380. doi: 10.1186/s13054-015-1097-0. PMID 26521922
- [Background] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Background] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498